CLINICAL TRIAL: NCT05365282
Title: Association Between Radial Artery Intervention and Development of Neuropathy in the Hand - A Prospective Study - The ACCESS IV Study
Brief Title: Association Between Radial Artery Intervention and Development of Neuropathy in the Hand - A Prospective Study
Acronym: ACCESS-IV
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Christian Juhl Terkelsen, Professor, Professor, Chief Physician, PhD., Aarhus University Hospital Skejby
Other Study IDs: 1-10-72-177-20
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Heart Disease; Nerve Injury; Carpal Tunnel Syndrome
Keywords: Transradial access; Ischemic Heart Disease; Hand Dysfunction
MeSH Terms: conditions — Myocardial Ischemia; Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Access pathway a. radialis (right or left) and neurophysiological measurements of the same hand (ipsilateral intervention group).
- Group B: Access pathway a.radialis (right or left) and neurophysiological measurements of opposite hand (contralateral intervention group).

SUMMARY:
Evaluation of potential nerve damage after radial CAG/PCI.

DETAILED DESCRIPTION:
Prospective patients scheduled for radial CAG/ PCI will be enrolled in the study. Prior to the procedure, sensory and motor nerve examination is performed at the wrists in both arms / hands. The examination is performed on both the median nerve and the ulnar nerve. Each patient acts as their own control. The nerve test is repeated bilaterally 1 month after the procedure. This creates 2 groups, A and B.

Patients will be asked to complete 2 questionnaires in relation to hand and arm symptoms. The patients ability to perform certain activities before and after the CAG/PCI procedure are also addressed. In addition, a diagnostic tool (Katz chart) will be completed, also before and after the CAG/PCI procedure.

Hypothesis:

Radial access is associated with an increased risk of pain and an increased incidence of nerve damage similar to the median nerve at the carpal tunnel or the ulnar nerve at the Guyon's canal.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be able to give informed consent

Exclusion Criteria:

* Pregnancy
* Negative Barbeau test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suspected of ischemic heart disease scheduled for radial CAG/PCI at Aarhus University Hospital
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological measurements | Aprox 1 hour
  The primary aim is the incidence/presence of electrofysiological signs of median and/or ulnar nerve lesion at the wrist and the presence of carpaltunnel syndrom.
  The electrodiagnosis of carpaltunnelsyndrom will be determined from the clinical picture and signs of prolonged distal motor lantency and reduced motor and sensory nerveconduction velocity across the wrist and/or reduced amplitudes of the median nerve and normal ulnar nerve at the wrist.

SECONDARY OUTCOMES:
Severity of hand symptoms and hand dysfunction | 10min
  Boston questionaire
Severity of hand symptoms and hand dysfunction | 10 min
  QuickDash questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Christian J Terkelsen, Professor, Study Chair — Aarhus University Hospital
Locations (1):
- Department of cardiology, Aarhus University Hospital in Skejby, Aarhus, Denmark